CLINICAL TRIAL: NCT03914560
Title: Evaluation of Macronutrients and Micronutrients Intakes in Burn Patients Treated as Outpatients
Brief Title: Nutritional Intakes in Burn Patients Treated as Outpatients
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Rousseau, Head of Clinic, Principal investigator, University of Liege
Other Study IDs: ABA
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Burns; Nutritional Deficiency
MeSH Terms: conditions — Burns; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Burn injury — minor burn injury

SUMMARY:
Nutrition is a key component of burn care. The primary goal of nutrition is to provide adequate supply in macro and micronutrients that are necessary to maintain organ function but also to wound healing, infection control and muscle preservation.

Studies about nutrition and burn care are mainly focused on severe burn patients. There is a few or no data regarding nutrition in minor burns. Those patients rarely receive a multidisciplinary approach, at least in Belgium.

The present study aimed to describe the nutritional condition of less severe burn patients treated as outpatients in a Belgian burn center. The ultimate goal was to determine whether this population needs specific dietetics follow-up or not.

ELIGIBILITY:
Inclusion Criteria:

* Burn treated exclusively in an outpatient clinic

Exclusion Criteria:

* Not french speaking
* Psychiatric disorders
* Patient refusal

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All burn patients admitted in the outpatient clinic of the investigator's burn center for minor burns
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
nutritional intakes | During the first week following injury
  Using a standardized food questionnaire, mean daily nutritional intakes were calculated for each patient (macronutrients and micronutrients). Food questionnaire is a questionnaire created by our dietetics unit, aiming to quantify the amount of food eaten at each meal. Quantities of macronutrients and micronutrients at each meal were then calculated using tables of food content (Nubel for all nutrients, excepting vitamin E calculated according Ciqual table).

SECONDARY OUTCOMES:
Body composition | During the first week following injury
  Body composition measured using bio impedance
Handgrip strength | During the first week following injury
  Strength measured an handheld dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Li§ge, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No